CLINICAL TRIAL: NCT02782637
Title: Prenatal Counseling in Extreme Prematurity: Parents' View
Acronym: PreCo-parents
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); UMC Utrecht (Other); Leiden University Medical Center (Other); Erasmus Medical Center (Other); Maastricht universitair medisch centrum, Maastricht (Unknown); Isala (Other); University Medical Center Groningen (Other); Maxima Medical Center (Other); Amsterdam UMC, location VUmc (Other); Fonds NutsOhra (Other)
Responsible Party: Sponsor
Other Study IDs: Preco-2
Record Dates: First submitted 2016-05-10; First posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Extreme Prematurity; Complications
Keywords: limits of viability; Prenatal Counseling; Decision-making; Viability; Counseling
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Survey and interviews: *part one* (quantitative)
  Survey on:
  A. prenatal counseling at the limits of viability, within three domains of interest:
  * organization of prenatal counseling
  * content of prenatal counseling
  * decision-making in prenatal counseling Domains used to evaluate current counseling and counseling preferences
  B. decision-making at the limits of viability: evaluation of the made decision (decisional conflict and regret)
  *part two* (qualitative)
  Individual interviews (qualitative) to in-depth explore preferences in prenatal counseling
  * insight in the specific preferred content of prenatal counseling.
  * study influencing factors on preferences in the domains of organization and decision-making.
  Interventions: Other: survey and interview

INTERVENTIONS:
Other: survey and interview — all participants: survey on prenatal counseling and treatment decisions at the limits of viability.
  a selection of participants: individual interviews to further perform in-depth exploration of prenatal counseling preferences

SUMMARY:
This study is part of the PreCo study, evaluating Dutch care in (imminent) extreme preterm birth including current and preferred counseling, barriers and facilitators for preferred counseling from both obstetricians and neonatologists, as well as parents' views on this.

Since 2010, intensive care can be offered in the Netherlands at 24+0 weeks gestation (with parental consent) but as some international guidelines, the Dutch guideline lacks detailed recommendations on organization, content and preferred decision-making of the counselling.

DETAILED DESCRIPTION:
The anticipated delivery of an infant at the limits of viability presents parents and professionals with medical, ethical and emotional issues; especially when a decision on the initiation of care has to be made. Since the first publication in 2002 by the American Academy of Pediatrics several (albeit different) guidelines and recommendations on periviability counseling have been published. However, there is no universally accepted way of performing prenatal counseling and, consequently, studies describe heterogeneous counseling practices worldwide.

Some guidelines on resuscitation at the limits of viability include recommendations on the parental involvement in the decision-making. Nevertheless, the extent of involvement and the gestational age (GA) at which parents should be involved varies. In 2010, the Dutch guideline on perinatal practice in extremely premature delivery lowered the limit offering intensive care from 25+0 to 24+0 weeks GA. Just as some international guidelines include a role for parents at the limits of viability, the Dutch guideline states that at 24 weeks GA informed consent of parents is required when initiating intensive care28. Although the guideline acknowledges the importance of prenatal counseling, recommendations on organization, content or decision-making of the counseling are very limited.

Although recommendations on counseling do exist, they may not be generally applicable in the Netherlands since cross-cultural differences in perinatal practices, healthcare organization, and physician and patient views are likely to exist. To compose a national framework on prenatal counseling at the limits of viability, the nationwide PreCo study (Prenatal Counseling in Prematurity) was designed, examining both professional and parental views. High quality of care originates when no differences exist between preferred and current counseling with uniformity between the involved caregivers (obstetricians and neonatologists) and specified to the needs of those receiving counseling, being the parents The PreCo study amongst parents has three major aims

1. to find initial preferences among Dutch experienced parents on prenatal counseling at the limits of viability (quantitatively)
2. to evaluate decision-making among Dutch experienced parents at the limits of viability (quantitatively)
3. to perform in-depth exploration of counseling preferences amongst Dutch parents (qualitatively)

ELIGIBILITY:
Inclusion Criteria:

* The study population consists of the cohort 01-10-2010 to 01-10-2013 of parents who were confronted with the birth of an extremely preterm infant with a gestational age between 24 and 25 weeks, after the introduction of the new Dutch guideline in October 2010.

Exclusion Criteria:

* birth at 24-25 weeks of gestation due to active termination of pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of the cohort 01-10-2010 to 01-10-2013 of parents who were confronted with the birth of an extremely preterm infant with a gestational age between 24 and 25 weeks, after the introduction of the new Dutch guideline in October 2010.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
current and preferred prenatal counseling practices in 3 domains (organization, content, decision-making) | during the time of the survey (march 2015 - march 2016)
evaluation of the decision made (decisional conflict and regret) | during the time of the survey (march 2015 - march 2016)
qualitative explored specific preferences in content, influencing factors on organization and decision-making | during the interviews (may - june 2015)

CONTACTS AND LOCATIONS:
Overall Officials: Marije Hogeveen, MD, PhD, Principal Investigator — Radboud